CLINICAL TRIAL: NCT00350766
Title: Multicenter Prospective Randomized Double Blind Trial of Bone Marrow Mononuclear Cells Transplantation Through Intracoronary Injection in Patients With Acute Myocardial Infarction.
Brief Title: Cell Therapy in Myocardial Infarction
Acronym: EMRTCC
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow recruitment rate and consequent financial exhaustion.
Sponsor: Ministry of Health, Brazil (Other Government)
Collaborators: Pro-Cardiaco Hospital (Other); Hospital do Coracao (Other); Instituto Estadual de Cardiologia Aloysio de Castro (Unknown); Hospital Cardiológico Costantini (Unknown); Hospital Universitário Regional do Norte do Paraná - FUEL (Unknown); Hospital Santa Izabel (Other); Hospital Santa Izabel de Sergipe (Unknown); Hospital Agamenon (Unknown); Hospital do Andaraí (Unknown); Hospital de Messejana (Unknown); Hospital de Clinicas de Porto Alegre (Other); Faculty of Medicine of Ribeirão Preto (FMRP-USP) (Other); Instituto Nacional de Cardiologia de Laranjeiras (Other); Instituto de Cardiologia do Rio Grande do Sul (Other); Hospital São Marcos (Unknown); Hospital Universitário Oswaldo Cruz - UPE (Unknown); Real Hospital Português de Beneficência (Unknown); Hospital Municipal Miguel Couto (Other); Anis Rassi Hospital, Brazil (Other); Federal University of São Paulo (Other); Instituto Dante Pazzanese de Cardiologia (Other); Universidade Federal do Rio de Janeiro (Other); Hospital Bandeirantes (Other); InCor Heart Institute (Other); Hospital Santa Isabel de Blumenau (Unknown); Federal University of Uberlandia (Other); Hospital TotalCor (Other); Hospital de Clínicas Mario Lioni (Unknown); Hospital de Clínicas de Niteroi (Unknown)
Responsible Party: Principal Investigator, Hans Fernando Rocha Dohmann, MD, PhD, Pro-Cardiaco Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMRTCC-IAM
Record Dates: First submitted 2006-07-10; First posted 2006-07-11 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Acute Myocardial Infarction
Keywords: Myocardial Infarction; Myocardial Ischemia; Ventricular Remodeling; Bone Marrow Cell Transplantation; Stem cells
MeSH Terms: conditions — Myocardial Infarction; Myocardial Ischemia; Ventricular Remodeling | interventions — Transplantation

STUDY DESIGN:
Intervention Model Description: Double Blind Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Control group received injection of saline with 5% autologous serum without the suspension of mononuclear cells.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated Group (Experimental): Intracoronary injection in the infarcted-related artery of 100 million bone marrow mononuclear cells resuspended in a 10 ml solution of saline with autologous serum.
  Interventions: Procedure: Autologous Bone Marrow Mononuclear Cells (ABMMC) Transplantation
- Control Group (Placebo Comparator): Intracoronary injection in the infarcted-related artery of placebo solution consisting of a saline containing autologous blood serum.
  Interventions: Procedure: Autologous Bone Marrow Mononuclear Cells (ABMMC) Transplantation

INTERVENTIONS:
Procedure: Autologous Bone Marrow Mononuclear Cells (ABMMC) Transplantation — Catheter based stem cells delivery of 100 million cells resuspended in a 10 ml solution of saline with autologous serum. About 100 ml of Bone Marrow aspirate were harvested from iliac crest between the fifth and seventh day after myocardial infarction. ABMMC were isolated by density gradient centrifugation on Ficoll-PaqueTM plus (Amersham Biosciences) and manipulated under aseptic conditions for injection, after being filtered through 100 um nylon mesh to remove cell aggregates.
  Other Names: Catheter based stem cell delivery

SUMMARY:
The purpose of this study is to determine cell therapy efficacy in patients with ST elevation acute myocardial infarction (STEMI)

DETAILED DESCRIPTION:
This study protocol describes a randomized double blind clinical trial, which main purpose is to evaluate the effect of the autologous bone marrow mononuclear cell (ABMMC) implant in 300 Brazilian patients with ST elevation acute myocardial infarction (STEMI).

Double blind study design was chosen for this trial, based on several phase I and II safety trials of intracoronary autologous bone marrow stem cells transplantation, already published. The study coordinator committee, supported by the Brazilian Health Ministry, therefore has proposed a phase III trial with the purpose of proving the efficacy of this kind of therapy, for a population with a high risk of developing heart failure and of death by cardiovascular cause.

Thus, in this protocol we propose a prospective, double blind, controlled and randomized trial to evaluate the effect of ABMMC transplantation through intracoronary infusion, on systolic left ventricle (LV) function. The main hypothesis of this trial is that patients submitted to autologous bone marrow stem cell implant, after 6 months follow up, will present a 5% relative increase of the ejection fraction (EF) comparing to control group.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be eligible if presenting all characteristics described below:

  * ST segment elevation myocardial infarction in two or more contiguous leads, and according to the WHO definition, at least one of the following two:

    i) Presence of chest pain. ii) Elevation of the myonecrosis markers.
  * Age between 30 and 80 years old.
  * Ejection fraction ≤50% on Echocardiogram (Simpson) and segmentary dysfunction of the infarction area, measured between the 3rd and 5th day post AMI.

Among patients submitted to thrombolytic therapy, the angioplasty of the related artery should be preferably done up to 24h after thrombolysis, with a maximum deadline of 72h after thrombolysis.

Exclusion Criteria:

* Patients will be ineligible if presenting any of the characteristics described below:

  * AMI related artery presenting TIMI < 3 at the moment f cell injection.
  * Left Main Coronary Artery Lesion of >50% or multivessel coronariopathy (>70% lesion in vessels with >2,0mm diameter in left anterior descending, circumflex and right coronary territory) indicating the need for CABG or angioplasty with three or more stents implant.
  * Coronary anatomy, after thrombolytic reperfusion, presenting no need for angioplasty with stent implant.
  * Final Diastolic Pression of the LV higher than 30 mmHg during ventriculography for evaluating EF inclusion criteria for the research protocol (item "c" of inclusion criteria).
  * Cardiac arrest or Killip IV AMI at admission with need of ventilatory support.
  * Cardiogenic shock persisting up to the third day after AMI (with need of Intra-aortic balloon pump or vasopressors).
  * AMI mechanical complications (ventricular septal defect, papillary muscle rupture, and left ventricular free wall rupture).
  * Significant valve disease, defined as aortic stenosis (mean systolic pressure gradient across the aortic valve >50mmHg), mitral stenosis with a valvar area less than 1,5 cm,2 moderate to severe aortic and/or mitral regurgitation.
  * Chronic use of immunosuppressive agents.
  * > 2,0 mg/dl creatinine or previous dialysis treatment.
  * Presence of fever on the past 48h before injection glaring active systemic infection according to ACCP/SCCM (American College of Chest Physicians/Society of Critical Care Medicine) sepsis definition.
  * Sustained ventricular tachycardia 48h after AMI.
  * Illicit drugs abuse or alcohol abuse (based on DSM IV).
  * Any co morbidity, with survival impact in two years.
  * Myocarditis
  * Active liver disease
  * COPD in continuous steroids use.
  * Hematological disease, neoplasm, bone disease or hemostatic disturbances.
  * Inflammatory disease or chronicle infectious disease.
  * Presence of definitive implantation of a cardiac pace maker or cardiac defibrillator.
  * Impossibility to reach a cells suspension of 100 million mononuclear cells due to cells paucity in the bone marrow aspirate.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2006-07-01 (Actual); Primary Completion 2014-01-21 (Actual); Study Completion 2014-07-14 (Actual)

PRIMARY OUTCOMES:
Global Left Ventricular Ejection Fraction change | 6 months

SECONDARY OUTCOMES:
Death | 30 days, 90 days, 6 months and 1 year
Acute myocardial infarction, stroke and hospital admission due to cardiovascular cause | 30 days, 90 days, 6 months and 1 year
Reintervention of the AMI related artery and of the non-related artery | 30 days, 90 days, 6 months and 1 year
Regional wall motion, wall thickening, and volume of late contrast enhancement | Baseline and 6 months
Evolutive alterations of the coronarian anatomy, as well as the patency of the coronary stents | 6 months
Quality of life assessment using the Short-Form 36, Minnesota Living with Heart Failure Questionnaire and Seattle Angina questionnaire | Baseline, 6 months and 1 year
Cost-effectiveness and cost-utility evaluation of autologous bone marrow mononuclear cells implant versus conventional treatment | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hans F Dohmann, MD, Principal Investigator — PROCEP/Pró-Cardíaco Hospital
Locations (1):
- PROCEP/Hospital Pró-Cardíaco, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dohmann HF, Silva SA, Sousa AL, Braga AM, Branco RV, Haddad AF, Oliveira MA, Moreira RC, Tuche FA, Peixoto CM, Tura BR, Borojevic R, Ribeiro JP, Nicolau JC, Nobrega AC, Carvalho AC. Multicenter double blind trial of autologous bone marrow mononuclear cell transplantation through intracoronary injection post acute myocardium infarction - MiHeart/AMI study. Trials. 2008 Jul 3;9:41. doi: 10.1186/1745-6215-9-41. PMID 18598362
- [Background] Tura BR, Martino HF, Gowdak LH, dos Santos RR, Dohmann HF, Krieger JE, Feitosa G, Vilas-Boas F, Oliveira SA, Silva SA, Bozza AZ, Borojevic R, de Carvalho AC. Multicenter randomized trial of cell therapy in cardiopathies - MiHeart Study. Trials. 2007 Jan 18;8:2. doi: 10.1186/1745-6215-8-2. PMID 17233910